CLINICAL TRIAL: NCT03772912
Title: Registry for the Use of HEMOBLAST Bellows in Total Knee Arthroplasty
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ETC 2018-006
Record Dates: First submitted 2018-12-06; First posted 2018-12-12 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Hemostatics; Coagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Total Knee Arthroplasty Patients: Patients undergoing primary or revision total knee arthroplasty procedures in which the surgeon elects to use HEMOBLAST Bellows to control minimal, mild, or moderate bleeding for which conventional means of hemostasis are ineffective or impractical
  Interventions: Device: HEMOBLAST Bellows

INTERVENTIONS:
Device: HEMOBLAST Bellows — The HEMOBLAST™ Bellows hemostatic agent consists of a bellows pre-loaded with 1.65g of powder composed of collagen, chondroitin sulfate, and thrombin (1500 IU). HEMOBLAST™ Bellows is indicated in surgical procedures as an adjunct to hemostasis when control of minimal, mild, and moderate bleeding by conventional procedures is ineffective or impractical, except in neurosurgical, ophthalmic, and urological procedures.

SUMMARY:
The purpose of this post-market observational registry is to collect additional data on the safety and effectiveness of the HEMOBLAST™ Bellows device in total knee arthroplasty procedures.

DETAILED DESCRIPTION:
A maximum of 100 subjects will be enrolled at up to 5 centers in the United States.

Enrollment occurs intraoperatively after confirmation of eligibility criteria. Data collection will occur during the surgical procedure as well as during patient follow up and will follow site standard of care. Subjects will be discontinued from the study after completion of the final follow up visit. The estimated duration of the study is approximately 10 months from the time of first subject enrollment to completion of the last subject follow up.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Patient is undergoing a unilateral total knee arthroplasty procedure; and
* Patient is willing and able to give written informed consent for registry participation.

Preoperative Exclusion Criteria:

* Patient has a known sensitivity or allergy to bovine and/or porcine substance(s); and
* Patient has religious or other objections to porcine, bovine, or human components.

Intraoperative Inclusion Criteria

* Patient has at least one Target Bleeding Site (TBS) with minimal, mild, or moderate bleeding for which conventional means for hemostasis are ineffective or impractical; and
* The surgeon elects to utilize HEMOBLAST™ Bellows per its approved Indication for Use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing elective, unilateral total knee arthroplasty procedures that meet all eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Achievement of Hemostasis at the Target Bleeding Site | Intraoperatively, expected within 3-10 minutes of application
  The ability of HEMOBLAST Bellows to achieve hemostasis (i.e. cessation of bleeding) at the target bleeding site will be assessed

SECONDARY OUTCOMES:
Incidence of Serious Adverse Device Effects (SADEs) | Through study completion, on average 1-2 days post-surgery
  The incidence of Serious Adverse Events deemed possibly, probably, or definitely related to the device will be quantified
Incidence of Unanticipated Serious Adverse Device Effects (UADEs) | Through study completion, on average 1-2 days post-surgery
  The incidence of Serious Adverse Events that are both unanticipated and deemed by the investigator to be possibly, probably, or definitely related to the device

IPD SHARING:
Plan to Share IPD: No